CLINICAL TRIAL: NCT06460961
Title: A Phase 1 Open-label, Multicenter Study of MK-6837 as Monotherapy and Combination Therapy in Participants With Advanced/Metastatic Solid Tumors
Brief Title: A Study of MK-6837 as a Monotherapy and Combination Therapy in Participants With Advanced/Metastatic Solid Tumors (MK-6837-001)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6837-001; MK-6837-001 (Other: MSD)
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Neoplasm Metastasis
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Cell Death 1 Ligand 1 (PDL1, PD-L1); Programmed Cell Death 1 Ligand 2 (PDL2, PD-L2)
MeSH Terms: conditions — Neoplasm Metastasis; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: MK-6837 Monotherapy (Experimental): Participants receive escalating doses of MK-6837 via intravenous (IV) infusion once every 3 weeks (Q3W) (Day 1 of every 21-day cycle) until progressive disease or discontinuation.
  Interventions: Biological: MK-6837; Drug: Rescue Medications
- Arm 2: MK-6837 + Pembrolizumab Combination Therapy (Experimental): Participants receive escalating doses of MK-6837 via IV infusion Q3W (Day 1 of every 21-day cycle) until progressive disease or discontinuation PLUS 200mg of pembrolizumab via IV infusion Q3W (Day 1 of every 21-day cycle) for up to 35 administrations (up to ~2 years).
  Interventions: Biological: MK-6837; Biological: Pembrolizumab; Drug: Rescue Medications

INTERVENTIONS:
Biological: MK-6837 — IV Infusion
Biological: Pembrolizumab — IV Infusion
  Other Names: MK-3475; KEYTRUDA®
  Arms: Arm 2: MK-6837 + Pembrolizumab Combination Therapy
Drug: Rescue Medications — Antihistamine, H2 receptor antagonist, acetaminophen (or equivalent), dexamethasone (or equivalent) administered per product label prior to MK-6837.

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and preliminary efficacy of MK-6837, administered as a monotherapy and in combination with pembrolizumab (MK-3475), in participants with histologically or cytologically confirmed advanced/metastatic solid tumors that have not responded to conventional therapy. There will not be any hypothesis testing in the study.

As of Amendment 04 (effective date: 18-Dec-2025), there are no pharmacokinetic (PK) secondary outcome measures in this study.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Histologically or cytologically confirmed solid tumor by pathology report that is advanced or metastatic
* Human Immunodeficiency Virus (HIV)-infected participants must have well controlled HIV on Antiretroviral Therapy (ART)
* Participants who are Hepatitis B Surface Antigen (HBsAg) positive are eligible if they have received Hepatitis B Virus (HBV) antiviral therapy for at least 4 weeks, and have undetectable HBV viral load before allocation
* Participants with history of Hepatitis C Virus (HCV) infection are eligible if HCV viral load is undetectable at screening

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Has not recovered to Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 or better from any Adverse Events (AEs) that were due to cancer therapeutics administered more than 4 weeks earlier
* History of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 2 years
* Has clinically significant cardiovascular disease
* HIV-infected participants with a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease
* Received prior systemic anticancer therapy including investigational agents within 4 weeks before the first dose of study intervention
* Has received any prior immunotherapy and was discontinued from that treatment due to a Grade 3 or higher immune-related AE (except endocrine disorders that can be treated with replacement therapy) or was discontinued from that treatment due to Grade 2 myocarditis or recurrent Grade 2 pneumonitis
* Received prior radiotherapy within 2 weeks of start of study intervention, or has radiation-related toxicities, requiring corticosteroids
* Received a live or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines is allowed
* Diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days before the first dose of study intervention
* Known additional malignancy that is progressing or has required active treatment within the past 2 years
* Known active Central Nervous System (CNS) metastases and/or carcinomatous meningitis
* Active autoimmune disease that has required systemic treatment in the past 2 years except replacement therapy
* History of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Active infection requiring systemic therapy
* History of allogeneic tissue/solid organ transplant
* Participants who have not adequately recovered from major surgery or have ongoing surgical complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2024-07-14 (Actual); Primary Completion 2027-07-13 (Estimated); Study Completion 2027-07-13 (Estimated)

PRIMARY OUTCOMES:
Number of participants who experience one or more dose-limiting toxicities (DLTs) | Cycle 1 (Up to approximately 21 days); each cycle is 21 days.
  The following events will be considered a DLT unless clearly due to underlying disease or extraneous causes: Grade 4 neutropenia lasting >7 days; Grade 3 or higher thrombocytopenia associated with clinically significant bleeding, regardless of duration; All Grade 3 or higher nonhematologic toxicities (with exceptions); Any abnormality that results in a drug induced liver injury; Febrile neutropenia Grade 3 or 4; Prolonged delay (>2 weeks) in initiating treatment after the first 21 days due to intervention-related toxicity; Any intervention-related toxicity that causes the participant to discontinue intervention during the first 21 days; Grade 5 toxicity. The number of participants who experience a DLT will be presented.
Number of participants who experience one or more adverse events (AEs) | Up to approximately 35 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Number of participants who discontinue study intervention due to an AE | Up to approximately 35 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (7):
- United States (3):
  - Atlantic Health System Morristown Medical Center ( Site 4001), Morristown, New Jersey
  - Providence Portland Medical Center ( Site 4002), Portland, Oregon
  - South Texas Accelerated Research Therapeutics (START) ( Site 4003), San Antonio, Texas
- Australia (2):
  - Westmead Hospital ( Site 1002), Westmead, New South Wales
  - The Alfred Hospital ( Site 1001), Melbourne, Victoria
- Princess Margaret Cancer Centre ( Site 2001), Toronto, Ontario, Canada
- Sheba Medical Center-ONCOLOGY ( Site 3001), Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/